CLINICAL TRIAL: NCT07372612
Title: A Prospective Randomized Controlled Trial of Flow-diverting Devices for the Treatment of Middle Cerebral Artery Bifurcation Aneurysms
Brief Title: Flow-diverting Devices for the Treatment of Middle Cerebral Artery Bifurcation Aneurysms
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, 庄宗, Deputy chief physician of Neurosurgery, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LCYJ-MS-11
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Aneurysms; Flow Diverter; Middle Cerebral Artery Aneurysm; Coiling Therapy
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flow diverter treatment group (Experimental): Flow diverter（FD, preferentially a Lattice stent) placement, with adjunctive minimal coiling of the aneurysm sac as needed.
  Interventions: Procedure: Flow diverter
- Stent-assisted coiling treatment group (Active Comparator): Underwent conventional stent-assisted coiling (preferentially using an LVIS stent)
  Interventions: Procedure: Stent-assisted coiling

INTERVENTIONS:
Procedure: Flow diverter — Flow diverter (FD, preferentially a Lattice stent) placement, with adjunctive minimal coiling of the aneurysm sac as needed
  Arms: Flow diverter treatment group
Procedure: Stent-assisted coiling — Conventional stent-assisted coil embolization was performed (with preferential use of an LVIS stent)
  Arms: Stent-assisted coiling treatment group

SUMMARY:
The goal of this clinical trial is to learn if flow diverter (FD) offers advantages over conventional stent-assisted coiling in the treatment of middle cerebral artery (MCA) bifurcation aneurysms . It will also learn about the safety of flow diverter (FD) treatment. The main questions it aims to answer are:

Does flow diverter (FD) treatment improves the rate of complete aneurysm occlusion and patients' neurological function? Does flow diverter (FD) treatment loweres the probability of aneurysm recurrence and the occurrence of complications?

Researchers will compare FD to a conventional stent-assisted coiling to see if FD treatment works better to treat MCA bifurcation aneurysms.

Participants will:

Undergo stent-assisted coiling or flow diverter treatment Take pre-operative and pre-discharge head MRI scans, neurological function assessments, and cognitive function assessments Visit the clinic 1 year for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Unruptured wide-necked middle cerebral artery bifurcation aneurysms definitively diagnosed by CTA or DSA;
2. Aneurysms requiring stent-assisted embolization with the necessity of preserving branch arteries;
3. Indication for either flow diversion device or conventional stent-assisted coiling;
4. Age between 18 and 70 years, inclusive;
5. The subject or their legally authorized representative has signed the written informed consent form.

Exclusion Criteria:

1. Concomitant significant organ dysfunction (e.g., severe cardiac, hepatic, or renal insufficiency), chronic inflammatory disease, or malignancy;
2. Pregnant or lactating women;
3. Presence of significant neurological deficit (mRS score > 2);
4. Presence of contraindications to flow diversion device or stent-assisted coiling (e.g., severe allergy to metallic material, contraindication to antiplatelet medication);
5. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Complete occlusion rate of middle cerebral artery bifurcation aneurysms at 1-year follow-up (assessed according to the Raymond-Roy Classification) | 1 year

SECONDARY OUTCOMES:
The rate of aneurysm recurrence at 1-year post-procedure | 1 year
Patients' neurological outcomes at 6 months and 1 year post-procedure (mRS scores and Mini-mental state examination) | 1 year
  The modified Rankin Scale (mRS) measures the degree of disability or dependence in the daily activities of patients. A score of 0 indicates no symptoms at all, score of 1 indicates no significant disability despite symptoms, score of 2 indicates slight disability, score of 3 indicates moderate disability, score of 4 indicates moderately severe disability, score of 5 indicates severe disability, and score of 6 indicates death.
Patients' cognitive outcomes at 6 months and 1 year post-procedure (MMSE scores) | 1 year
  The Mini-mental state examination（MMSE） examination includes time and place orientation, registration,attention and calculation, recall, language,repitition, complex commands. Score excess 24 or more indicates a normal cognition, 19-23 points indicates mild cognitive impairment, score of 10-18 points indicates moderate cognitive impairment and score below 9 points indicates severe cognitive impairment
Incidence of Branch Vessel Patency and In-stent Stenosis Assessed by Digital Subtraction Angiography (DSA) | 1 year
  Branch vessel patency (specifically the covered M2 branches) will be evaluated using follow-up DSA images and classified as patent, narrowed, or occluded. In-stent stenosis is defined as a narrowing of the vessel diameter >50% within the stented segment compared to the reference vessel diameter.
Total interventional procedure time (from puncture to completion of the procedure) | 1 year

IPD SHARING:
Plan to Share IPD: No